CLINICAL TRIAL: NCT07332832
Title: Evaluation of Suspicious Prostate Lesions Via Sequential Bi-parametric MRI: A Multi-center Prospective Cohort Study
Brief Title: Sequential bpMRI for Suspicious Prostate Lesions
Acronym: SEQ-bpMRI
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Collaborators: Shanghai East Hospital of Tongji University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025R0590
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; Magnetic resonance imaging; Follow up
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Prostate biopsy tissue for pathological diagnosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MRI follow-up cohort of patients with clinically suspected prostate cancer: Scheduled Follow-up: All enrolled patients will undergo a follow-up period of 24 months. Every 6 months: PSA testing, Digital Rectal Examination (DRE), and clinical assessment. At months 12 and 24: Repeat bi-parametric MRI (bpMRI) examinations.
  Biopsy Decision-Making:
  Triggered Biopsy: During the follow-up period (e.g., at month 12), a prostate biopsy will be recommended if the patient exhibits MRI progression to PI-RADS 4/5, or presents with PI-RADS 3 combined with a PSA density (PSAD) > 0.2 ng/ml².
  Endpoint Biopsy: To ensure study rigor and safety, patients who have not undergone biopsy due to radiological progression during the 24-month follow-up will be advised to undergo a confirmatory biopsy at the study endpoint (month 24). This aims to maximally exclude the missed diagnosis of clinically significant prostate cancer (csPCa).
  Interventions: Diagnostic Test: PSA test; Diagnostic Test: Bi parametric MRI

INTERVENTIONS:
Diagnostic Test: PSA test — Blood PSA test every 6 months
Diagnostic Test: Bi parametric MRI — Bi parametric MRI examination every year.

SUMMARY:
This study aims to establish a prospective exploratory cohort and database to observe the dynamic evolution of bi-parametric MRI (bpMRI). We intend to investigate the clinical utility of sequential MRI combined with prostate biopsy in the diagnosis of prostate cancer. Specifically, by utilizing bpMRI findings and their dynamic changes to guide the timing of biopsies, we aim to avoid unnecessary procedures. Furthermore, the safety and efficacy of this strategy will be assessed through long-term follow-up, ultimately promoting the precision diagnosis and treatment of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 85 years.
* Total PSA (tPSA) level ranging from 3 ng/ml to 20 ng/ml (inclusive).
* Underwent prostate MRI at the study institution with complete imaging sequences.
* Capable of providing written informed consent.
* Patients with PI-RADS 4-5, or PI-RADS 3 combined with PSAD ≥ 0.2 ng/ml², who have undergone prostate biopsy with no diagnosis of clinically significant prostate cancer (csPCa).
* Biopsy-naïve patients with PI-RADS 2, or PI-RADS 3 combined with PSAD < 0.2 ng/ml².

Exclusion Criteria:

* Pathologically confirmed diagnosis of clinically significant prostate cancer (csPCa).
* Contraindications to prostate biopsy or inability to tolerate the procedure.
* Current use of 5-alpha reductase inhibitors (5-ARIs).
* History of hip replacement, metallic hip arthroplasty, or extensive pelvic orthopedic surgery with metallic hardware, or presence of other implants that would degrade MRI image quality.
* Contraindications to bi-parametric MRI (bpMRI) (e.g., severe claustrophobia, cardiac pacemakers).

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical suspicion of prostate cancer presenting to Peking University First Hospital and Shanghai East Hospital (Affiliated to Tongji University)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
csPCa detection rate | From enrollment to the end of follow up at 24 weeks
  Clinically significant prostate cancer detection rates across different radiological changes (progression, stability, and regression)

IPD SHARING:
Plan to Share IPD: Undecided